CLINICAL TRIAL: NCT03758963
Title: A Prospective, Multi-center, Randomized, Double-blinded (Subject & Independent Efficacy Evaluator), Comparative Clinical Study to Evaluate the Efficacy and Safety of SRT (Selective Retina Therapy) With 'R:GEN' in Patients With Central Serous Chorioretinopathy
Brief Title: Selective Retina Therapy With 'R:GEN' in Patients With Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTN-02
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, double-blinding will be applied for subjects and independent efficacy evaluators. It is difficult to apply blinding to the practitioner who handles the products used for therapy because of difference in the procedure of the treatment and sham, but the information related to the medical device shall not be released to subjects and independent efficacy evaluators. For blinding of independent efficacy evaluators, an independent evaluator shall conduct efficacy evaluation tests (OCT, BCVA test, contrast sensitivity test, FA).
  Subjects and independent efficacy evaluators will not know which group the subjects are assigned to and whether SRT or sham procedure is used. The blinding on the test device will be maintained until the data for statistical analysis are opened.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Laser (Experimental): 1. Once the energy to be applied for the treatment is determined through the laser irradiation testing, conduct laser therapy after selecting "T" corresponding to treatment laser on GUI.
  2. At irradiation, excluding the circle area with a 100 μm radius (200 μm diameter) from the center of the fovea, irradiate laser in the form of surrounding the leakage site with an interval of 0.5-1 spot diameter (fovea = 1 spot size). As for the test spots, the serial number needs to be given for each treatment spot with the order of irradiation, as described above.
  3. If pigment epithelial detachment (PED) occurs at the leakage site, irradiate laser around the PED (excluding the circle area with a 100 μm radius (200 μm diameter) from the center), not to the leakage site.
  4. Within 2 hours after therapy, perform tests for efficacy evaluation (color fundus photography and fluorescein angiography).
  Interventions: Device: R:GEN Selective Retina Therapy
- Sham Laser procedure (Sham Comparator): 1. Select "C" corresponding to Sham Therapy on GUI of the laser device, and then perform Sham therapy.
     * During Sham therapy, for patient's blinding, both light from the slit lamp and sound from laser oscillation are same as laser irradiation, and no laser oscillation will occur for treatment.
  2. Perform subsequent procedures in the same manner as the procedure of study group.
  Interventions: Device: R:GEN Selective Retina Therapy

INTERVENTIONS:
Device: R:GEN Selective Retina Therapy — Selective Retina Therapy (SRT) is the treatment method using innovative laser technology with the wavelength absorbed by melanosomes such as laser photocoagulation, but due to short pulse width (1.7 µs) with 100 Hz repetition rate, Retinal Pigment Epithelium (RPE) cells may be destroyed only through the generation of microbubble around melanosomes (photomechanical action), and no thermal damage of normal cells or tissues may occur in the surrounding tissues. SRT influences the RPE wound healing, including migration and proliferation of RPE cells, which treats CSC in the mechanism of recovering RPE. Once RPE is recovered, the sub-retinal fluid may be pumped out and retinal function again recovered. Moreover, previous studies showed that SRT may stimulate a moderate increase of activated metalloproteinase (MMP), leading to the improvement of Bruch's membrane's transport property.

SUMMARY:
The purpose of this clinical study is to evaluate the efficacy and safety of selective retina therapy (SRT) using R:GEN, an approved laser device, in patients with central serous chorioretinopathy.

DETAILED DESCRIPTION:
In this study, treatment effect of each group will be evaluated by follow-up once a month of both study group and control group other than the 2nd month until 6 months following the first procedure.

For the primary efficacy evaluation, the percentage of subjects who show complete removal of sub-retinal fluid (SRF) in Optical Coherence Tomography (OCT) results will be evaluated in the study group, before SRF therapy and at 3 months after therapy, and in control group, before sham procedure using R:GEN and at 3 months after therapy. In addition, for secondary efficacy evaluation, major symptoms of central serous chorioretinopathy will be evaluated at 3 and 6 months including changes in best corrected visual acuity (BCVA) on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart, the degree of retinal functional damage, and changes in sub-retinal fluid (SRF) and central macula thickness (CMT) on OCT. At 6 months, removal rate of leakage on Fluorescene Angiography (FA) and recurrence of the disease will be evaluated to compare the recurrence rate of study group and control group undergoing sham procedure.

The subjects in the study group who only meet the conditions of retreatment at 3 ~ 5 months after selective retina therapy (SRT) may receive SRT up to twice again.

The subjects in the control group those who have not recovered naturally but have persistent clinical symptoms at 3 months will undergo SRT. And the subjects in the control group who only meet the conditions of retreatment at 5 months after SRT at 2 months.

And the subjects in the control group, who have experienced complete disappearance of SRF at 3 months after Sham procedure, but SRF is observed again at 4 or 5 months, may receive SRT up to twice again.

These subjects will be categorized into a separate subgroup and the efficacy and safety of SRT will be evaluated every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult patients aged 19 or over and less than 55
2. Patients who have had clinical symptoms of central serous chorioretinopathy over 3 months.
3. Patients whose best corrected visual acuity (BCVA) is at least 20/200 based on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart (BCVA based on the ETDRS chart will be converted into logMAR)
4. Patients with Sub-Retinal Fluid (SRF) that has been going into the fovea continuously
5. Patients with ≥1 ~ ≤ 3 active leakage sites in Fundus Fluorescein Angiography (FA)
6. Patients who are of child-bearing potential and have agreed to use a medically acceptable contraceptive method during the study period

   ☞Medically acceptable contraceptive method: Condom, oral contraceptive pills that have been continued for more than three months, contraceptive injection or implants or intrauterine contraceptive device
7. Patients who voluntarily agree to participate in this study, and are willing to and able to follow the protocol.

Exclusion Criteria:

1. Patients with other retinal diseases such as choroidal neovascularization, polypoidal choroidal vasculopathy.
2. Patients with the conditions that make laser therapy difficult such as cataract or vitreous cloudiness.
3. Patients who have atrophy (diameter: ≥1000㎛) in the retinal pigment epithelium including the fovea.
4. Patients who had undergone laser or photodynamic therapy for central serous chorioretinopathy prior to the study participation.
5. Patients who have received steroid treatment (periocular, subtenon, intraocular) within the last one year
6. Patients who have received intraocular injection of anti-Vascular Endothelial Growth Factor (anti-VEGF) agent within the last six months.
7. Patients who have undergone ophthalmological surgery such as intraocular surgery or vitrectomy within the last six months.
8. Patients who have taken medication for central serous chorioretinopathy such as acetazolamide, spironolactone, and kalidinogenase [within the last two months].
9. Patients who have a history of allergy to fluorescein used for FA and indocyanine green used for ICG angiography.
10. Female patients who are pregnant or breastfeeding.
11. Patients with systemic diseases such as Cushing's syndrome, inflammatory diseases, uncontrolled hypertension and diabetes, liver diseases, kidney diseases.
12. Patients who have pigment epithelial detachment that is directly related to the point of leakage with a diameter of more than 1000 μm.
13. Patients who are considered ineligible for this study according to the investigator's judgment.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Sub-retinal Fluid (SRF) Removal Rate | 3 months
  The percentage of subjects (%) who show complete removal of Sub-retinal Fluid (SRF) on Optical Coherence Tomography (OCT) is compared between study group and control group.

SECONDARY OUTCOMES:
Improvement of Best Corrected Visual Acuity | 3, 6 months
  The improvement of Best Corrected Visual Acuity is evaluated using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart and is compared between study group and control group.
Degree of Retinal Functional Damage | 3, 6 months
  The degree of retinal functional damage is compared between study group and control group.
Change in Sub-retinal Fluid (SRF) | 3, 6 months
  The change in Sub-retinal Fluid (SRF) (μm, mm3) on Optical Coherence Tomography (OCT) is compared between study group and control group.
Change in Central Macular Thickness | 3, 6 months
  The change on Central Macular Thickness (CMT) (μm) based on Optical Coherence Tomography (OCT) results are compared between the study and control group.
Removal Rate of Leakage | 6 months
  The percentage (%) of participants who show complete removal of leakage in Fluorescene Angiography (FA) results is compared between study group and control group.
Recurrence Rate | 6 months
  The percentage (%) of participants who show recurrence is compared between study group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Oh Woong Kwon, PhD, Principal Investigator — Nune Eye Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam hospital, Seoul
  - Nune Eye Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul ST.Mary's Hospital, Seoul
  - The Catholic University of Korea Yeouido St.Mary's Hospital, Seoul